CLINICAL TRIAL: NCT07108075
Title: Acute Portal Pressure Reduction by Metformin and Carvedilol Compared to Carvedilol Alone in Cirrhosis - a Randomised, Double Blind Study.
Brief Title: Acute Portal Pressure Reduction by Metformin and Carvedilol Compared to Carvedilol Alone in Cirrhosis.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ILBS-ACLF-25
Record Dates: First submitted 2025-07-15; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis | interventions — Carvedilol; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metformin and Carvedilol (Experimental): Metformin (1000 mg) Carvedilol (12.5 mg)
  Interventions: Drug: Carvedilol; Drug: Metformin
- Carvedilol (Active Comparator): Carvedilol (12.5 mg)
  Interventions: Drug: Carvedilol

INTERVENTIONS:
Drug: Carvedilol — Carvedilol 12. 5mg
Drug: Metformin — Metformin 1000 mg
  Arms: Metformin and Carvedilol

SUMMARY:
Clinically significant portal hypertension (CSPH) is defined as HVPG >10 mmHg. Patients with CSPH are at risk of developing esophageal varices and clinical decompensation (variceal bleeding, ascites, jaundice, encephalopathy), which mark the transition from compensated stage to a stage of the disease (decompensated) associated with higher mortality (1). HVPG is calculated by subtracting the free hepatic venous pressure (FHVP), a measure of systemic pressure, from the wedged hepatic venous pressure (WHVP), a measure of hepatic sinusoidal pressure. HVPG is surrogate marker in many clinical applications such as gold standard test to evaluate presence and severity of portal hypertension (PHT) diagnosis, risk stratification, monitoring of the patients on beta blockers (2). Non selective beta-blockers like propranolol and carvedilol are indicated in adults for primary and secondary prophylaxis of variceal hemorrhage. Acute hemodynamic response to intravenous propranolol with HVPG values coming down to <12 mm Hg or reduction to >20% from baseline have been shown to be associated with reduced long term risk of variceal bleed. Metformin has also recently showed to reduce portal pressure in a randomised control study. The mechanism of action of metformin is different from beta blockers (by increasing nitric oxide by upregulating iNOS and eNOS). Hence we are planning the current work to evaluate Acute portal pressure reduction by Metformin and Carvedilol compared to Carvedilol alone in cirrhosis - a randomised, double blind study.

ELIGIBILITY:
Inclusion Criteria:

- Consecutive patients of cirrhosis with variceal bleed.

Exclusion Criteria:

1. Age < 18 and > 75yr,
2. CTP Score ≥12,
3. Patients of cirrhosis without variceal bleed,
4. Patients on metformin, nonselective β-blockers or carvedilol treatment within last 5 days,
5. S.Bilirubin > 3 mg/dl,
6. S.creatinine 1.5 mg/dl,
7. Contraindications to NSBB (heart rate < 60 /min, BP < 110/60 mm Hg,
8. Asthma, heart failure),
9. PVT,
10. HCC
11. HE grades 2-4

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-06-14 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
HVPG response (decrease by ≥ 20 % from baseline or < 12 mmHg). | 2 hours

SECONDARY OUTCOMES:
HVPG decrease by ≥ 10% in both groups. | 2 hours
Reduction in HVPG in both groups. | 2 hours
Change in blood sugar level after 2 hours of the drug in both groups. | 2 hours
Change in inflammatory markers (IL-10, TNF α, i-NOS, e-NOS) in both groups. | 2 hours
Change in liver and spleen stiffness. | 2 hours
Change in cardiac output in both groups. | 2 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences (ILBS), New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided